CLINICAL TRIAL: NCT01642069
Title: Observational - NUP98/JARID1A as a Recurrent Aberration in Pediatric Acute Megakaryoblastic Leukemia
Brief Title: Studying Genes in Samples From Younger Patients With Acute Megakaryoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B9; NCI-2012-01984 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-15; First posted 2012-07-17 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Myeloid Leukemia/Other Myeloid Malignancies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Cryopreserved specimens are analyzed for NUP98 fusion to NSD1, JARID1A, and TOP1, myeloid/lymphoid or MLL-rearrangements, and other gene expression profiling by RT-PCR and karyotyping or FISH. Results are then compared with each patient's outcome data.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is looking into genes in samples from younger patients with acute megakaryoblastic leukemia (AMKL). Studying samples of blood, tissue, and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in RNA and identify biomarkers related to cancer

DETAILED DESCRIPTION:
Study Subtype: Ancillary/Correlative Observational Study Model: Cohort Time Perspective: Retrospective Biospecimen Retention: Samples With DNA Biospecimen Description: Cryopreserved mRNA Study Population Description: Samples from AAML0531 Sampling Method: Non-Probability Sample

OBJECTIVES:

I. To determine whether NUP98/JARID1A expression is a recurrent translocation in NUP98-rearranged cases in pediatric acute megakaryoblastic leukemia (AMKL).

II. To screen the Children Oncology Group (COG) samples for genetic aberrations in pediatric AMKL.

OUTLINE:

Cryopreserved specimens are analyzed for NUP98 fusion to NSD1, JARID1A, and TOP1, myeloid/lymphoid or mixed-lineage leukemia (MLL)-rearrangements, and other gene expression profiling by reverse transcriptase polymerase chain reaction (RT-PCR) and karyotyping or fluorescence in situ hybridization (FISH). Results are then compared with each patient's outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Cryopreserved specimens of pediatric patients diagnosed with acute megakaryoblastic leukemia

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with acute megakaryoblastic leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR, defined as less than 5% blasts in the bone marrow, with regeneration of tri-lineage hematopoiesis, plus absence of leukemic cells in the cerebrospinal fluid or elsewhere) | Up to 8 weeks
Probability of event-free survival (pEFS, defined as time between diagnosis and first event, including non-remitting, death of any cause and second malignancy) | Up to 8 weeks
Overall survival (pOS, defined as time between diagnosis and death) | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soheil Meshinchi, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States